CLINICAL TRIAL: NCT02478762
Title: Reevaluation of the Glycemic Objectives of Women With Gestational Diabetes Mellitus
Brief Title: Glycemic Objectives of Women With Gestational Diabetes Mellitus
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: very difficult recruitment
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Principal Investigator, Jean-Luc Ardilouze, Endocrinologist, Université de Sherbrooke
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14-160
Record Dates: First submitted 2015-06-16; First posted 2015-06-23 (Estimated); Last update posted 2018-05-03 (Actual); Status verified 2018-05

CONDITIONS: Gestational Diabetes Mellitus
Keywords: Foetal glycated hemoglobin; Glycemic objectives treatment
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Normal glycemic control (Active Comparator): GDM women in this group will reach glycemic objectives recommended by the Canadian Diabetes Association: fasting: 5.3 mmol/L and 2-hour after meals: 6.7 mmol/L.
  Interventions: Procedure: Normal glycemic control
- Low glycemic control (Experimental): GDM women in this group will reach lower glycemic objectives than those recommended by the Canadian Diabetes Association: fasting: 4.8 mmol/L and 2-hour after meals: 5.9 mmol/L.
  Interventions: Procedure: Low glycemic control

INTERVENTIONS:
Procedure: Normal glycemic control — Use diet, physical exercise of insulins to reach normal glycemic control.
  Arms: Normal glycemic control
Procedure: Low glycemic control — Use diet, physical exercise of insulins to reach low glycemic control.
  Arms: Low glycemic control

SUMMARY:
In a previous study, the investigators established the dosage of foetal glycated hemoglobin (FGH). It represents the mean of blood sugar 4-6 before the delivery. The investigators also compared the FGH of newborn of women with and without gestational diabetes mellitus (GDM) and determined that newborn of women with GDM had significantly higher FGH that newborn of women without GDM.

In this study, the investigators want to compare the FGH of newborn of GDM women randomized to a group reaching the Canadian Diabetes Association recommended blood glucose objectives treatment (fasting: 5.3 mmol/L and 2-hour after meals: 6.7 mmol/L) to a group reaching lower blood glucose objectives (fasting: 4.8 mmol/L and 2-hour after meals: 5.9 mmol/L)

ELIGIBILITY:
Inclusion Criteria:

* gestational age between 15 and 32 weeks since last menstrual date,
* received education on gestational diabetes mellitus,
* able to read and understand French.

Exclusion Criteria:

* known type 1 or type 2 diabetes,
* treatment interfering woth glucose metabolism,
* deficit may hinder the understanding of the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2015-03; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Foetal glycated hemoglobin | At delivery

SECONDARY OUTCOMES:
Treatment satisfaction | End of pregnancy
  Evaluated by questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Luc Ardilouze, MD, PhD, Principal Investigator — Université de Sherbrooke
Locations (1):
- Centre de recherche du Centre hospitalier universitaire de Sherbrooke, Sherbrooke, Quebec, Canada